CLINICAL TRIAL: NCT03294915
Title: Effect of Resistant Starch From Green Banana Flour on the Insulin Sensitivity of Subjects With Prediabetes: Randomized Clinical Trial
Brief Title: Effect of Resistant Starch on Insulin Sensitivity and Beta Cell Function in Subjects With Prediabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-0155
Record Dates: First submitted 2017-06-28; First posted 2017-09-27 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2017-09

CONDITIONS: Prediabetes
Keywords: prediabetes; resistant starch; insulin sensitivity
MeSH Terms: conditions — Prediabetic State; Insulin Resistance | interventions — Resistant Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistant Starch (Active Comparator): Green banana flour
  Interventions: Dietary Supplement: Resistant Starch
- Placebo (Placebo Comparator): Maltodextrin, cellulose and guar gum
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Resistant Starch — Addition of 42g per day of green banana flour (10g / day resistant starch) to the usual diet of study participants
  Arms: Resistant Starch
Dietary Supplement: Placebo — Addition of 42g per day of mixture of guar gum, maltodextrin and cellulose to the usual diet of study participants
  Arms: Placebo

SUMMARY:
To compare the use supplementation based on green banana flour versus placebo in the insulin sensitivity on individuals who have prediabetes.

DETAILED DESCRIPTION:
In order to evaluate whether supplementation with green banana flour may improve insulin sensitivity of individuals with prediabetes, volunteers will be recruited by advertising on the web page of Hospital de Clinical de Porto Alegre. After screening and selection, they will be submitted to a clinical, laboratory and nutritional standard evaluation, assessment of physical activity and body fat composition.The laboratory evaluation will include the oral glucose tolerance test (OGGT 75g), lipid profile, insulin, C-peptide, glycated hemoglobin and glycated albumin. Insulin sensitivity and beta-cell function will be assessed by the hyperglycemic CLAMP before and after the intervention.Interim statistical analysis will be performed at the end of the participation of ten study volunteers.

Subjects will receive green banana flour or placebo for four weeks.

ELIGIBILITY:
Inclusion criteria

1. Serum glycated hemoglobin (A1c) values between 5.7 and 6.5%, or fasting glucose ≥ 5.55 mmol/L and < 6.94 mmol/L or oral glucose tolerance test (75g) ≥7.77 and <11.04 mmol /L.
2. Body mass index (BMI) ≥ 25 kg / m² (≥23 kg / m² for those of Asian origin) and ≤ 35 kg / m² for screening.
3. Stable weight (maximum variation of approximately 5%) for at least 4 weeks prior to screening.
4. Apt and willing to provide the written informed consent term and to comply with the requirements of the study protocol.

Exclusion Criteria:

1. Clinically symptomatic gastrointestinal disease including, but not limited to, inflammatory bowel disease.
2. History of gastric bypass, antrectomy, or resection of the small intestine.
3. History of chronic pancreatitis or acute idiopathic pancreatitis.
4. Myocardial infarction, coronary artery bypass grafting, post-transplant cardiomyopathy or stroke in the last 6 months.
5. Any anomaly in clinical laboratory tests which may prevent safe participation in the study.
6. Tumor diagnosed and / or treated (except basal cell skin cancer, cervical carcinoma in situ, or prostate cancer in situ) within the past 5 years.
7. Hemoglobinopathy or chronic anemia known.
8. Donation of one unit (500 ml) or more of blood, significant loss of blood equivalent to at least one unit of blood within the last 2 weeks or blood transfusion in the last 8 weeks.
9. Any concomitant medical condition / disorder which, in the investigator's opinion, is likely to:

   * Will interfere with the patient's ability to complete the entire study period or participate in all study activities;
   * Require, during the study, the administration of a treatment that may affect the interpretation of the efficacy and safety data.
10. Treatment with any oral antidiabetic medicinal product and / or herbal preparations / non-prescription medicines that may affect glycemic control within 12 weeks prior to screening.
11. Chronic treatment with oral or parenteral corticosteroids (> 7 consecutive days of treatment) within 4 weeks prior to screening.
12. Treatment with weight-reducing agents (eg, orlistat, sibutramine, topiramate, bupropion) within the last 12 weeks prior to screening.
13. History of unstable hypertension (> 170/105 mmHg) in the last 12 weeks prior to screening.
14. Treatment with a lipid-lowering drug that has not been kept in a stable dose within the last 8 weeks prior to screening.
15. Treatment with thyroid hormone that has not been kept in a stable dose in the last 12 weeks prior to screening.
16. Investigational drug use within 30 days or 5 half-lives (whichever is longer) prior to screening unless guidelines from local health authorities require a longer period.
17. Any of the following laboratory abnormalities in screening:

    * Alanine aminotransferase (ALT) and / or Aspartate aminotransferase (AST) 3 times the upper limit of normality;
    * Glomerular filtration estimated by the equation kidney disease ≤ 60 ml per min by 1.73 m².
    * Fasting triglycerides > 5.6 mmol / L;
    * Thyroid stimulating hormone (TSH) outside normal range.
18. History of substance abuse (including alcohol) within the last year.
19. Women with potential to become pregnant and / or who are using local or systemic hormonal contraceptive method; Women in the follicular phase of the menstrual cycle and also pregnant and lactating women.
20. Potentially unreliable patients and those considered by the Investigator as unsuitable for the study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity | 4 weeks
  Insulin sensitivity compared to the baseline visit measured by hyperglycemia clamp

SECONDARY OUTCOMES:
Hormonal changes | 4 weeks
  Alteration of hormones that affect glucose metabolism, such as peptide C
Change in lipid profile | 4 weeks
  Alteration of total cholesterol, HDL-cholesterol and triglycerides
Change total body fat | 4 weeks
  Change total body fat will be compared before and after the intervention by means of bioimpedance
Beta cell function | 4 weeks
  Beta cell function (first and second phase of insulin secretion) will be measured by hyperglycemic clamp
Glycemic control | 4 weeks
  Measured by hemoglobin glycated

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Gerchman, MD, Principal Investigator — Federal University of Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahn SE, Prigeon RL, McCulloch DK, Boyko EJ, Bergman RN, Schwartz MW, Neifing JL, Ward WK, Beard JC, Palmer JP, et al. Quantification of the relationship between insulin sensitivity and beta-cell function in human subjects. Evidence for a hyperbolic function. Diabetes. 1993 Nov;42(11):1663-72. doi: 10.2337/diab.42.11.1663. PMID 8405710
- [Background] Johnston KL, Thomas EL, Bell JD, Frost GS, Robertson MD. Resistant starch improves insulin sensitivity in metabolic syndrome. Diabet Med. 2010 Apr;27(4):391-7. doi: 10.1111/j.1464-5491.2010.02923.x. PMID 20536509
- [Background] Asp NG, van Amelsvoort JM, Hautvast JG. Nutritional implications of resistant starch. Nutr Res Rev. 1996 Jan;9(1):1-31. doi: 10.1079/NRR19960004. No abstract available. PMID 19094263
- [Background] Higgins JA. Resistant starch: metabolic effects and potential health benefits. J AOAC Int. 2004 May-Jun;87(3):761-8. PMID 15287677
- [Background] Maki KC, Carson ML, Miller MP, Turowski M, Bell M, Wilder DM, Reeves MS. High-viscosity hydroxypropylmethylcellulose blunts postprandial glucose and insulin responses. Diabetes Care. 2007 May;30(5):1039-43. doi: 10.2337/dc06-2344. Epub 2007 Jan 26. PMID 17259476
- [Background] Moulin CC, Tiskievicz F, Zelmanovitz T, de Oliveira J, Azevedo MJ, Gross JL. Use of weighed diet records in the evaluation of diets with different protein contents in patients with type 2 diabetes. Am J Clin Nutr. 1998 May;67(5):853-7. doi: 10.1093/ajcn/67.5.853. PMID 9583841
- [Background] Kahn SE, Hull RL, Utzschneider KM. Mechanisms linking obesity to insulin resistance and type 2 diabetes. Nature. 2006 Dec 14;444(7121):840-6. doi: 10.1038/nature05482. PMID 17167471
- [Background] Kahn SE, Zraika S, Utzschneider KM, Hull RL. The beta cell lesion in type 2 diabetes: there has to be a primary functional abnormality. Diabetologia. 2009 Jun;52(6):1003-12. doi: 10.1007/s00125-009-1321-z. Epub 2009 Mar 27. PMID 19326096
- [Background] Perreault L, Pan Q, Mather KJ, Watson KE, Hamman RF, Kahn SE; Diabetes Prevention Program Research Group. Effect of regression from prediabetes to normal glucose regulation on long-term reduction in diabetes risk: results from the Diabetes Prevention Program Outcomes Study. Lancet. 2012 Jun 16;379(9833):2243-51. doi: 10.1016/S0140-6736(12)60525-X. Epub 2012 Jun 9. PMID 22683134
- [Background] Tabak AG, Herder C, Rathmann W, Brunner EJ, Kivimaki M. Prediabetes: a high-risk state for diabetes development. Lancet. 2012 Jun 16;379(9833):2279-90. doi: 10.1016/S0140-6736(12)60283-9. Epub 2012 Jun 9. PMID 22683128
- [Background] Englyst HN, Kingman SM, Cummings JH. Classification and measurement of nutritionally important starch fractions. Eur J Clin Nutr. 1992 Oct;46 Suppl 2:S33-50. PMID 1330528
- [Background] Murphy MM, Douglass JS, Birkett A. Resistant starch intakes in the United States. J Am Diet Assoc. 2008 Jan;108(1):67-78. doi: 10.1016/j.jada.2007.10.012. PMID 18155991
- [Background] Robertson MD, Wright JW, Loizon E, Debard C, Vidal H, Shojaee-Moradie F, Russell-Jones D, Umpleby AM. Insulin-sensitizing effects on muscle and adipose tissue after dietary fiber intake in men and women with metabolic syndrome. J Clin Endocrinol Metab. 2012 Sep;97(9):3326-32. doi: 10.1210/jc.2012-1513. Epub 2012 Jun 28. PMID 22745235
- [Background] DeFronzo RA, Tobin JD, Andres R. Glucose clamp technique: a method for quantifying insulin secretion and resistance. Am J Physiol. 1979 Sep;237(3):E214-23. doi: 10.1152/ajpendo.1979.237.3.E214. PMID 382871
- [Background] Sjaarda L, Lee S, Tfayli H, Bacha F, Bertolet M, Arslanian S. Measuring beta-cell function relative to insulin sensitivity in youth: does the hyperglycemic clamp suffice? Diabetes Care. 2013 Jun;36(6):1607-12. doi: 10.2337/dc12-1508. Epub 2012 Dec 28. PMID 23275361
- [Background] Tarini J, Wolever TM. The fermentable fibre inulin increases postprandial serum short-chain fatty acids and reduces free-fatty acids and ghrelin in healthy subjects. Appl Physiol Nutr Metab. 2010 Feb;35(1):9-16. doi: 10.1139/H09-119. PMID 20130660
- [Background] Anderson JW, Davidson MH, Blonde L, Brown WV, Howard WJ, Ginsberg H, Allgood LD, Weingand KW. Long-term cholesterol-lowering effects of psyllium as an adjunct to diet therapy in the treatment of hypercholesterolemia. Am J Clin Nutr. 2000 Jun;71(6):1433-8. doi: 10.1093/ajcn/71.6.1433. PMID 10837282
- [Background] Menezes EW, Tadini CC, Tribess TB, Zuleta A, Binaghi J, Pak N, Vera G, Dan MC, Bertolini AC, Cordenunsi BR, Lajolo FM. Chemical composition and nutritional value of unripe banana flour (Musa acuminata, var. Nanicao). Plant Foods Hum Nutr. 2011 Sep;66(3):231-7. doi: 10.1007/s11130-011-0238-0. PMID 21732181